CLINICAL TRIAL: NCT02471300
Title: Pilot Study to Evaluate the Effect of Fasting on the Asthma Inflammasome
Brief Title: Effect of Fasting on the Asthma Inflammasome
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150136; 15-H-0136
Record Dates: First submitted 2015-06-12; First posted 2015-06-15 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: Asthma; Inflammasome; Fasting; Airflow Obstruction
MeSH Terms: conditions — Asthma; Fasting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: stable mild-moderate asthmatic subjects

SUMMARY:
Background:

Research shows that restricting calories has a positive effect on immune cell health in healthy people. Researchers want to learn if it will help people with asthma. They want to better understand how the body s immune response and lung function responds to short-term calorie restriction. For this, they want people to fast (no food or drink except water) for 24 hours.

Objective:

To explore the benefits of calorie restriction in people with asthma.

Eligibility:

Healthy people ages 18 to 60 who have a history consistent with asthma and prior documentation of airflow obstruction or wheezing.

Design:

* Participants who have taken part in asthma research at NIH will be screened with a telephone interview. All other participants will have a medical history, blood tests, and physical exam.
* Eligible participants will return to the NIH Clinical Center one morning for 2 hours. They will be fed breakfast. They may have blood and urine tests.
* Participants will then fast for 24 hours.
* Participants will return to the Clinical Center the next morning for 4 hours. They will have blood drawn. They will eat breakfast and then repeat blood draws 2.5 hours later. They will have a urine test.
* Blood and urine tests will be done at the end of the fast and after the meals to confirm that the participant fasted for the full 24-hour period.
* Participants will have lung function tests and exhaled gas measurements. A machine will measure the volume of air they can breathe out. Some gases in the breath increase with inflammation. Participants will breathe into a machine that analyzes the gases in their breath.

DETAILED DESCRIPTION:
The NLRP3 inflammasome is part of the innate immune system that can be activated by atherosclerosis, gout and diabetes (sterile inflammation). As mitochondrial signaling can trigger the NLRP3 inflammasome, we initially proposed that fasting, via a nutrient-sensing mitochondrial program, would dampen this innate immune program. Our preliminary data shows that a 24-hour fasting does blunt NLRP3 inflammasome activation in healthy young individuals. Interestingly, this inflammasome program has been implicated in the pathophysiology of bronchoreactivity linked to asthma and intermittent fasting has been found to reduce disease exacerbations in asthmatic patients. The objective of this protocol will extend our investigations, from what we are finding in young control normal volunteers, to enable us to investigate stable mild-moderate asthmatic subjects to determine whether fasting can blunt inflammasome activation and assess whether this transient nutrient-deprivation maneuver can improve airflow. Blood samples and pulmonary function testing to assay the immune response and bronchoreactivity will be performed in subjects in response to a 24-hour fast (water intake will not be restricted) followed by re-testing 3 hours after a fixed caloric meal. The objective of this pilot study is to identify if these immune adaptive pathways can be subdued in human subjects with a known inflammasome linked disease. Additionally, this study may enable us to identify a potential therapeutic pathway to blunt/negate inflammation associated with nutrient-excess associated bronchoreactivity of asthma.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Males and females between the ages of 18 and 60
* Asthmatic subjects will have a history consistent with asthma, be on chronic asthma therapy and have prior documentation of reversible airflow obstruction based upon either a positive response to an inhaled bronchodilator or a positive methacholine bronchoprovocation challenge test

EXCLUSION CRITERIA:

* Subjects with concurrent acute illness or other chronic illnesses associated with inflammation including diabetes requiring medical management.
* Female subjects who are pregnant or lactating
* Subjects who have donated blood or participated in another clinical trial involving blood draws in the last 8 weeks.
* Medical condition identified by screening bloodwork that would preclude safe participation or valid data collection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: -Males and females between the ages of 18 and 60@@@-Asthmatic subjects will have a history consistent with asthma, be on chronic asthma therapy and have prior documentation of reversible airflow obstruction based upon either a positive response to an inhaled bronchodilator or a positive methacholine broncho-provocation challenge test@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-08-26 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Change in IL-1-beta secretion in response to inflammasome stimulation in PBMCs comparing the fasted response to the fed response | 24 hours
  Determine whether the NLRP3 inflammasome is blunted by a 24-hour fast in PBMC s in subjects with mild to moderate asthma.Initiate 24-hour fast with the exception of drinking water and use of asthma medications until midnight. Patients will be asked to hold their asthma medications after midnight. Fasting research labs to study the inflammasome and Fed State Research Labs to study the inflammasome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Sack, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Besnard AG, Guillou N, Tschopp J, Erard F, Couillin I, Iwakura Y, Quesniaux V, Ryffel B, Togbe D. NLRP3 inflammasome is required in murine asthma in the absence of aluminum adjuvant. Allergy. 2011 Aug;66(8):1047-57. doi: 10.1111/j.1398-9995.2011.02586.x. Epub 2011 Mar 28. PMID 21443539
- [Background] Kim SR, Kim DI, Kim SH, Lee H, Lee KS, Cho SH, Lee YC. NLRP3 inflammasome activation by mitochondrial ROS in bronchial epithelial cells is required for allergic inflammation. Cell Death Dis. 2014 Oct 30;5(10):e1498. doi: 10.1038/cddis.2014.460. PMID 25356867
- [Background] Kim HY, Lee HJ, Chang YJ, Pichavant M, Shore SA, Fitzgerald KA, Iwakura Y, Israel E, Bolger K, Faul J, DeKruyff RH, Umetsu DT. Interleukin-17-producing innate lymphoid cells and the NLRP3 inflammasome facilitate obesity-associated airway hyperreactivity. Nat Med. 2014 Jan;20(1):54-61. doi: 10.1038/nm.3423. Epub 2013 Dec 15. PMID 24336249
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-H-0136.html